CLINICAL TRIAL: NCT02740257
Title: Skin Lesion Detection With Novel Total Body Digital Photography Smartphone Application
Brief Title: Smartphone Application to Detect Skin Lesions
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Beatrice Nardone, Research Assistant Professor, Northwestern University
Other Study IDs: STU00202166
Record Dates: First submitted 2016-03-31; First posted 2016-04-15 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Skin Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 Artificial Lesions: Photos will be taken of skin lesion markings using a smartphone
  Interventions: Other: Photos
- Group 2 high risk: A convenience sample of patients will be recruited. This population will consist of patients with known high risk to have new/changing lesions, and who fall within the Fitzpatrick skin types I-IV. High risk patients include, but are not limited to, those with dysplastic nevus syndrome, previous history of melanoma/non-melanoma skin cancer, fair skin, >16 nevi, family history of melanoma, and/or immunosuppressed status. The first photography session will be taken by the research team in all 13 projections. After the first visit, the patient will be instructed to take photographs every month for 12 months using the TBDP app on their smart phone or tablet, and have follow-up research appointments every 6 months.
  Interventions: Other: Photos

INTERVENTIONS:
Other: Photos — Photos will be taken of skin lesion markings using a smart phone or tablet

SUMMARY:
The primary objective of Part One of this study is to determine the sensitivity of an automated total body digital photography (TBDP) app to detect color and size changes in the human skin, and whether a new lesion has arisen.

The primary objective of Part Two is to test the sensitivity and specificity as well as feasibility of field use of an automated TBDP app to detect pigmented and non-pigmented skin lesions in high risk populations.

DETAILED DESCRIPTION:
SkinIO is an early-stage healthcare IT company specializing in education, early detection, and prevention of skin cancer. This study will utilize their product, skinIO, an enhanced full-body skin cancer screening system that works on mobile devices and tablets to track changes in skin over time without any additional imaging hardware. skinIO enables dermatology staff to photograph high-risk patients in 13 medical photography poses to quickly capture full-body skin surfaces at multiple resolutions using a mobile device. These images are automatically uploaded to a HIPAA-compliant server environment where they will be rapidly processed to detect any spots, lesions, and moles. Dermatologists will then be able to annotate these images and flag specific images for follow-up every month.

In order to assess whether or not the software will accurately detect spot changes, the investigators will test the product on a sample of volunteer subjects.

Part One:

The study population will undergo one study visit. This visit will include 2 sets of photos taken by the research team after the collection of a small amount of identifying and contact information for each subject. There will be an initial 3-5 photographs taken of areas of the body that have at least 3 natural or artificial skin markings (ie. moles, angiomas, scars, keloids, seborrheic keratosis, small tattoos, etc). These markings will allow the app to calculate the parameters of any original lesions, and thereby more accurately detect new markings or changes based on these calculations. Once the original photographs are taken, one of each individual's original skin marking will be enhanced/enlarged with a marking pen, as well as 3- 5 new marks added to the skin. A Sharpie brush tip permanent marker will be utilized to make the new skin markings. These markers have been AP certified to be non-toxic. The following colors have been chosen: orange, black, brown, red, blue, purple, yellow and pink. A second photograph will be taken of the same areas of the body chosen for initial photographs to determine if the application could detect the changes. This group will not have their images sent to a dermatologist for evaluation, as they are artificially produced.

Part Two:

In order to test the sensitivity and feasibility of field of use of the TBDP app, a second convenience sample of patients will be recruited. Recruitment will be done in waiting rooms with the attending physician's consent. If needed, recruitment will be done outside of the waiting room in the form of flyers, website and e-mail announcements. This population will consist of patients with known high risk to have new/changing lesions, and who fall within the Fitzpatrick skin types I-IV. High risk patients include, but are not limited to, those with dysplastic nevus syndrome, previous history of melanoma/non-melanoma skin cancer, fair skin, >16 nevi, family history of melanoma, and/or immunosuppressed status. The first photography session will be taken by the research team in all 13 projections. Each projection corresponds to each body area that will be photographed to ensure total body photography. After the first visit, the patient will be instructed to take photographs every month for 12 months using the TBDP app on their smart phone or tablet, and have follow-up research appointments every 6 months. The patient will be provided a user guide with written instructions for application use. The TBDP app has a built-in reminder system for the patient. Any changes detected by the app will be stored on the research team's database. Standard of care will be followed for any new/changing lesions. Patients will be recommended to have a follow-up appointment with their dermatologist, within 2 weeks. No procedures will be completed by the research team, and a physician will not be seeing the patients during their research appointments. During these visits, the research team will compare the photographs taken by the TBDP app to the patient's skin to see how sensitive the app is. Patients will continue their regular office visits at 6 months and/or 12 months as per standard of care for high risk patients. The research team will use information from chart reviews for assessment of the outcome for new or changing lesions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 - 85.
* Subjects with the following skin types:

  1. Always burns, never tans or
  2. Burns easily, then develops light tan or
  3. Burns moderately, then develops light tan or
  4. Burns minimally rarely, then develops moderate tan.
* Subjects who deny prior skin reactions to washable markers.
* Subjects who have natural skin markings on at least 3 areas of their body.
* Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator in English.
* Subjects are able to complete the study procedures.
* Subjects are willing to have digital photos taken of them.

Exclusion Criteria:

* Subjects who have a history of skin disease (eg. vitiligo, psoriasis)
* Subjects with the following skin types:

  1. Never burns, always develops a dark tan or
  2. Never burns, no noticeable change in appearance.

Part Two (only):

H] Subjects must be high risk. High risk is defined as subjects with conditions including, but not limited to: dysplastic nevus syndrome, previous history of melanoma/non-melanoma skin cancer, fair skin, >16 nevi, family history of melanoma, immunosuppressed status I] Subjects must have an iPhone 4S or newer, or an iPad Air 2, iPad Mini 4 or iPad Pro in order to download and use the application and take photographs of high enough quality for the physician to analyze if needed.

J] Subjects must have someone who is able to take photos of the subject every month. The designated individual may or may not be present at the initial encounter.

4.2 Exclusion Criteria A] Subjects who have a history of skin disease (eg. vitiligo, psoriasis)

B] Subjects with the following skin types:

1. Never burns, always develops a dark tan or
2. Never burns, no noticeable change in appearance. Part Two (only) C] Subjects without the appropriate devices for app download. The appropriate devices are iPhone 4s or newer, or iPad Air 2, iPad Mini 4 or iPad Pro.

D] Subjects who do not have someone who is capable of taking photos of the subject every month.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with various skin types (Fitzpatrick I-IV)
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-03; Primary Completion 2018-11-07 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of an automated total body digital photography (TBDP) | Baseline
  We will assess whether or not the photography software can accurately detect spot changes. We will test the product on a sample of volunteer subjects. The study population will undergo one study visit and will include 2 sets of photos. There will be an initial 3-5 photographs taken of areas of the body that have at least 3 natural or artificial skin markings. These markings will allow the app to calculate the parameters of any original lesions, and thereby more accurately detect new markings or changes based on these calculations. Once the original photographs are taken, one of each individual's original skin marking will be enhanced/enlarged with a marking pen, as well as 3-5 new marks added to the skin. A Sharpie brush tip permanent marker will be utilized to make the new skin markings. A second photograph will be taken of the same areas of the body chosen for the initial photographs in order to determine if the application could detect the changes.

SECONDARY OUTCOMES:
Sensitivity of an automated total body digital photography (TBDP) in high risk subjects | Baseline, 6 and 12 months follow-up
  Data will be compared between the last picture taken by the app before the clinic visit and the lesions seen by the clinician at the clinic visit. Total number of lesions will be those detected by the clinician, which were not present in the baseline skin evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Nardone, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brewer AC, Endly DC, Henley J, Amir M, Sampson BP, Moreau JF, Dellavalle RP. Mobile applications in dermatology. JAMA Dermatol. 2013 Nov;149(11):1300-4. doi: 10.1001/jamadermatol.2013.5517. PMID 24067948
- [Result] Kohler BA, Sherman RL, Howlader N, Jemal A, Ryerson AB, Henry KA, Boscoe FP, Cronin KA, Lake A, Noone AM, Henley SJ, Eheman CR, Anderson RN, Penberthy L. Annual Report to the Nation on the Status of Cancer, 1975-2011, Featuring Incidence of Breast Cancer Subtypes by Race/Ethnicity, Poverty, and State. J Natl Cancer Inst. 2015 Mar 30;107(6):djv048. doi: 10.1093/jnci/djv048. Print 2015 Jun. PMID 25825511
- [Result] Suneja T, Smith ED, Chen GJ, Zipperstein KJ, Fleischer AB Jr, Feldman SR. Waiting times to see a dermatologist are perceived as too long by dermatologists: implications for the dermatology workforce. Arch Dermatol. 2001 Oct;137(10):1303-7. doi: 10.1001/archderm.137.10.1303. PMID 11594853
- [Result] Tsang MW, Resneck JS Jr. Even patients with changing moles face long dermatology appointment wait-times: a study of simulated patient calls to dermatologists. J Am Acad Dermatol. 2006 Jul;55(1):54-8. doi: 10.1016/j.jaad.2006.04.001. Epub 2006 May 6. PMID 16781292
- [Result] Jacobson CC, Resneck JS Jr, Kimball AB. Generational differences in practice patterns of dermatologists in the United States: implications for workforce planning. Arch Dermatol. 2004 Dec;140(12):1477-82. doi: 10.1001/archderm.140.12.1477. PMID 15611425
- [Result] Robson Y, Blackford S, Roberts D. Caution in melanoma risk analysis with smartphone application technology. Br J Dermatol. 2012 Sep;167(3):703-4. doi: 10.1111/j.1365-2133.2012.11046.x. Epub 2012 Jul 5. No abstract available. PMID 22762381
- [Result] Ferrero NA, Morrell DS, Burkhart CN. Skin scan: a demonstration of the need for FDA regulation of medical apps on iPhone. J Am Acad Dermatol. 2013 Mar;68(3):515-6. doi: 10.1016/j.jaad.2012.10.045. No abstract available. PMID 23394920
- [Result] Wolf JA, Moreau JF, Akilov O, Patton T, English JC 3rd, Ho J, Ferris LK. Diagnostic inaccuracy of smartphone applications for melanoma detection. JAMA Dermatol. 2013 Apr;149(4):422-6. doi: 10.1001/jamadermatol.2013.2382. PMID 23325302